CLINICAL TRIAL: NCT06922799
Title: A Comparison Between Orthodontic and Non-orthodontic Patients on Oral Indexes and Salivary pH and Quality: Cross-sectional Study
Brief Title: A Comparison Between Orthodontic and Non-orthodontic Patients on Oral Indexes and Salivary pH and Quality
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Other Study IDs: 2025-SALIVARYPH
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Dental Plaque; Saliva Altered
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Orthodontic group: Patients from this group are candidate to orthodontic treatment
  Interventions: Diagnostic Test: Saliva-Check Buffer test and periodontal charting
- Orthodontic group: Patients from this group are undergoing an orthodontic treatment
  Interventions: Diagnostic Test: Saliva-Check Buffer test and periodontal charting

INTERVENTIONS:
Diagnostic Test: Saliva-Check Buffer test and periodontal charting — Saliva-Check buffer test will be used to perform evaluations on saliva pH, quantity and quality

SUMMARY:
This study aims to assess the caries susceptibility in pediatric patients aged 6-14 years old using Saliva-Check Buffer salivary tests. A total of 40 patients will be enrolled, divided into two groups:

1. Group A (Pre-Orthodontic Treatment): this group will include pediatric patients who have completed dental treatments (mechanical debridement, fillings, extractions) and have not yet started orthodontic treatment.
2. Group B (Orthodontic Treatment): this group will consist of pediatric patients who have been undergoing orthodontic treatment for at least 6 months.

DETAILED DESCRIPTION:
This study aims to assess the caries susceptibility in pediatric patients aged 6-14 years old using Saliva-Check Buffer salivary tests. A total of 40 patients will be enrolled, divided into two groups:

1. Group A (Pre-Orthodontic Treatment): this group will include pediatric patients who have completed dental treatments (mechanical debridement, fillings, extractions) and have not yet started orthodontic treatment.
2. Group B (Orthodontic Treatment): this group will consist of pediatric patients who have been undergoing orthodontic treatment for at least 6 months.

Ethical Considerations: the study will be conducted in accordance with the Declaration of Helsinki and the norms of the Good Clinical Practice.

Patient Enrollment: patients meeting the inclusion criteria will be identified from the dental clinic's patient records. Parents or legal guardians will be approached to obtain informed consent for participation in the study.

Baseline Assessment: baseline dental examinations will be conducted to assess the dental health status of each patient, recording the following indexes: DMFT (Decayed, Missing, Filled Teeth), DMFS, PCR. Then, saliva collection and testing will be performed with Saliva-Check Buffer.

Data Analysis: data will be statistically analysed. Normality test will be performed, and a parametric or non-parametric test will be performed to compare the two groups for all the variables tested. Significance threshold will be predefined for p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients about to begin orthodontic treatment or already undergoing orthodontic therapy
* Willingness to undergo Saliva-Check Buffer salivary tests.
* Parental or legal guardian consent for participation in the study.

Exclusion Criteria:

* Patients with systemic medical conditions that may affect the results of salivary tests.
* Patients unwilling or unable to cooperate for saliva sample collection required for the tests.
* Patients who have taken antibiotics or other medications that could influence saliva composition in the weeks prior to testing.
* Patients with oral anomalies that may interfere with data collection or affect test results.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: Patients recruited from the Unit of Orthodontics and Pediatric Dentistry, Section of Dentistry, Department of Clinical, Surgical, Diagnostic and Pediatric Sciences, University of Pavia, Pavia, Italy
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-18 (Actual)

PRIMARY OUTCOMES:
DMFT (Decayed, Missing, Filled Teeth) | Baseline
  Sum of decayed, missing due to caries, and filled teeth.
DMFS (Decayed, Missing, Filled Surfaces) | Baseline
  Sum of decayed, missing due to caries, and filled tooth surfaces.
PCR (Plaque Control Record) | Baseline
  Number of surfaces with plaque / Total number of surfaces examined) x 100 using disclosing Tri Plaque ID gel.
Frankl Behavioral Scale | Baseline
  Classification of patients based on cooperation during treatment, using a scale from 1 to 4:
  * 1: Definitely positive Good rapport with the dentist, interested in the dental procedures, laughing and enjoying the situation.
  * 2: Positive Acceptance of treatment; at times cautious, willingness to comply with the dentist, at times with reservation but patient follows the dentist's directions cooperatively.
  * 3: Negative Reluctant to accept treatment; uncooperative, some evidence of negative attitude but not pronounced, i.e. /sullen, withdrawn.
  * 4: Definitely negative Refusal of treatment, crying forcefully, fearful or any other overt evidence of extreme negativism.
Saliva Check Buffer test | Baseline
  Complete assessment of saliva quality, quantity and pH

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator